CLINICAL TRIAL: NCT00962286
Title: Effect of Furosemide on Obesity-induced Glomerular Hyperfiltration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The blood pressure did not decrease following furosemide administration
Sponsor: Rabin Medical Center (Other)
Responsible Party: Boris Zingerman, MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBEFUR
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Obesity-induced Hyperfiltration
Keywords: Furosemide; obesity
MeSH Terms: conditions — Obesity | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Furosemide, obesity, glomerular hyperfiltration (Experimental)
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Subjects will receive 300 mg of lithium carbonate at 22.00 the day before the renal function tests.Intravenous catheters will be placed in each upper limb for infusion of clearance markers and blood sampling.A priming dose of inulin (50 mg/kg) and p-aminohippuric acid (8 mg/kg) will be administered. Thereafter, inulin and p-aminohippuric acid will be infused continuously. A 200-300 ml water load will be given during the first 60-min prime.
  Subjects will be started on furosemide p.o. 20 mg every 12 hours, starting on day 1 at 15.00 after the renal function studies. Nine doses will be taken, the last dose on day 4 at 7 am.
  In case the blood pressure does not decrease following 20 mg bid furosemide administration, the study will be repeated after 4 weeks using a dose of 40 mg p.o. bid.

SUMMARY:
Background: Obesity is associated with a high prevalence of chronic kidney disease. The glomerular hyperfiltration associated with obesity may play a role in the pathogenesis of obesity associated chronic kidney disease. Attenuation of hyperfiltration by pharmacological means may slow down the development and progression of chronic renal failure. The investigators have previously shown that acetazolamide, a proximally acting diuretic that activates TGF by increasing solute delivery to the macula densa, abates glomerular hyperfiltration. The present study was designed to test the hypothesis that this decrease in hyperfiltration is specific to acetazolamide and not due to a non specific diuretic effect. The aim of the present study is to evaluate the effects of the administration of furosemide p.o. to subjects with severe obesity on glomerular hemodynamics.

Methods: Ten obese subjects will participate in the study. They will undergo measurement of glomerular filtration rate (inulin clearance) (GFR), renal plasma flow (RPF) (p-aminohippuric acid clearance), filtration fraction, fractional excretion of lithium (FE LI) and blood pressure, before and after administration of oral furosemide 20 to 40 mg bid for 3 days. The effects of furosemide on glomerular hemodynamics in obese subjects will be compared to the previously studied effects of acetazolamide.

DETAILED DESCRIPTION:
Almost half of the causes of death in the industrial world are due to cardio-vascular disease. Two of the main risk factors for CV disease have become much more prevalent during the last decades, reaching epidemic dimensions in the 21st century: hypertension and obesity. In 2003-2004, 66% of the adult US population had a BMI over 25, while 32% had a BMI over 30 .Hypertension is more prevalent in obese than in lean subjects .The cause and effect relationship between these two conditions is supported by the fact that weight loss is associated with a decrease in blood pressure .

Salt retention by the kidney is one of the important mechanisms involved in the pathogenesis of hypertension in obesity. Studies in animal models and in humans showed that increased salt reabsorption occurs in the tubules in obesity . Another renal functional abnormality occurring in obesity is glomerular hyperfiltration, characterized by increased RPF and increased GFR up to twice the normal level . The structural basis to these functional abnormalities is renal hypertrophy and glomerular enlargement.

These functional and structural abnormalities have deleterious consequences:

1. Increased urinary albumin excretion. Microalbuminuria, an important risk factor for CV disease, has a high prevalence in obese subjects .
2. Increased risk for the development of focal segmental glomerulosclerosis, the so-called obesity related glomerulopathy. The incidence of this disease has multiplied 10 times within 15 yrs in the USA .
3. Increased rate of progression of chronic renal insufficiency in kidney disease not primarily caused by obesity. Following initial glomerular damage from any cause, the number of remnant functioning glomeruli decreases. The consequent compensatory increase in single nephron filtration rate of these remnant glomeruli leads to further glomerular damage in kidney disease not related to obesity . In the obese with chronic renal damage, the obesity related hyperfiltration amplifies the compensatory augmentation in single nephron GFR of remnant nephrons, thus worsening glomerular damage, irrespective of the cause of the primary insult.

The clinical relevance of these abnormalities is reflected in the sharp increase in the risk of developing end stage renal disease in the obese. This relative risk, independently of confounders as diabetes mellitus, hypertension and dyslipidemia, is 3 to 5 depending on the severity of obesity .

Considering the role of hyperfiltration in the pathogenesis of CKD in the obese, attenuation of hyperfiltration by pharmacological means may slow down the development and progression of chronic renal failure. One of the tools available is activating TGF. Tubuloglomerular feedback (TGF) refers to the alterations in GFR that can be induced by changes in tubular flow rate. An increase in the delivery of chloride to the macula densa results in a reduction in GFR, resulting in a decrease in the tubular flow rate delivered to the macula densa . An increase in chloride delivery to the macula densa can be obtained by administrating acetazolamide, a diuretic acting on the proximal tubule. We have previously shown that administration of acetazolamide to obese subjects results in attenuation of glomerular hyperfiltration.

The aim of the present study is to show that the effect of acetazolamide on GFR is specific and not due to its diuretic effect. We will study the effects of furosemide, a diuretic which does not activate TGF ,on GFR and RPF in obese subjects.

METHODS

Inclusion criteria:

10 obese men (BMI>30), aged 18 to 55, with glomerular hyperfiltration (creatinine clearance>130 ml/min) will be included in the study.

Exclusion criteria:

Any of the following conditions:

* Heart failure
* Known allergy to furosemide, inulin or amino-hippurate
* Pharmacologic treatment for hypertension, cardiac disease, diabetes mellitus
* Treatment with corticosteroids or NSAID

Methods:

A 24-hour urine collection will be performed during the week prior to the renal function test studies for assessment of sodium intake. Subjects will receive 300 mg of lithium carbonate at 22.00 the day before the renal function tests. They will be instructed to drink 250 ml of water at bedtime. Renal function tests will start at 08.00 a.m. after a 10-hour fast, excepting a drink of 250 ml of water at 07.00 a.m. Intravenous catheters will be placed in each upper limb for infusion of clearance markers and blood sampling. After blood sampling for urea, creatinine, proteins, glucose, electrolytes, blood gases, insulin, renin, aldosterone, Hba1c, CBC. A priming dose of inulin (50 mg/kg) and p-aminohippuric acid (8 mg/kg) will be administered. Thereafter, inulin and p-aminohippuric acid will be infused continuously. A 200-300 ml water load will be given during the first 60-min prime. Four accurately timed urine collections of 40-60 minutes will then be obtained by spontaneous voiding. Peripheral venous blood will be drawn to bracket each urine collection. Arterial pressure will be measured by a trained observer, after 30 minutes of rest in the supine position, using an electronic oscillometric blood pressure measuring device (Datascope, Accutorr). The cuff will be appropriately sized to the diameter of the arm and the arm positioned at the heart level. At least 4 measurements will be performed during the study, each measurement being the mean of 3 readings.

Subjects will be started on furosemide 20 mg every 12 hours, starting on day 1 at 15.00 after the renal function studies. Nine doses will be taken, the last dose on day 4 at 7 am.

In case the blood pressure does not decrease following 20 mg bid furosemide administration, the study will be repeated after 4 weeks using a dose of 40 mg bid.

Laboratory procedures: Plasma and urinary concentrations of inulin and p-aminohippuric acid will be analyzed by colorimetric methods (22,23). Lithium in serum and urine will be measured using the ICP-OES (Inductively Coupled Plasma Optical Emission Spectrometer) method. Urine microalbumin will be determined by competitive chemiluminescent enzyme immunoassay (Imulite, DPC, Los Angeles, CA, USA).

Calculations: GFR will be determined from the average value for the timed inulin clearances, and renal plasma flow (RPF) - from the average value for the timed p-aminohippurate clearances. The fractional excretion of lithium (FE Li) will be calculated as lithium clearance / GFR, using two timed urine collections. FE Li will be determined as the average value for these two measurements Statistical Analysis: The significance of differences between groups will be evaluated by paired and unpaired two-tailed Student's t-test. The Student's t-test will be applied to non-normally distributed data (albumin excretion rate and fractional lithium excretion) after log transformation. P<0.05 will be considered as significant. The response to treatment with furosemide will be compared to the previously studied response to treatment with acetazolamide.

ELIGIBILITY:
Inclusion Criteria:

* 10 obese men (BMI>30), aged 18 to 55, with glomerular hyperfiltration (creatinine clearance>130 ml/min) will be included in the study.

Exclusion Criteria:

* Any of the following conditions:

  * Heart failure
  * Known allergy to furosemide, inulin or amino-hippurate
  * Pharmacologic treatment for hypertension, cardiac disease, diabetes mellitus
  * Treatment with corticosteroids or NSAID

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
change in GFR | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Boris Zingerman, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] 1. Chagnac A et al: Glomerular hemodynamics in severe obesity. Am J Physiol Renal Physiol. 2000;278(5):F817-22. 2. Chagnac A et al: The effects of weight loss on renal function in patients with severe obesity. J Am Soc Nephrol. 2003 Jun;14(6):1480-6. 3. Navar LG: Renal autoregulation: perspectives from whole kidney and single nephron studies. Am J Physiol. 1978 May;234(5):F357-70. 4. Deng A etal: Hemodynamics of early tubuloglomerular feedback resetting during reduced proximal reabsorption. Kidney Int. 2002 Dec;62(6):2136-43. 5. Dupont AG et al: Renal pharmacodynamic effects of torasemide and furosemide in normal man.Drug Res. 38(1) 1a 1998 172-175.